CLINICAL TRIAL: NCT05163054
Title: Cohort Study of Patients With Type 1 Diabetes Registered With Mobile Application in China
Acronym: COOPERATIONS
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021380
Record Dates: First submitted 2021-11-09; First posted 2021-12-20 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2021-10

CONDITIONS: Type 1 Diabetes
Keywords: cohort study; type 1 diabetes; mobile; home-community-hospital; China
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Whole blood sample and urine sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
For last decade, the innovation of mobile health platform has brought new opportunities for disease management. Previous studies have shown that health management programs based on mobile platforms for patients with diabetes can improve patients' glucose control, self-management ability and quality of life. Type 1 diabetes mellitus (T1DM) due to its characteristics needs long-term linkage care throughout the lifespan cycle of patients. Therefore, this study intends to construct a prospective and open T1DM cohort based on mobile application and platform, to deliver home-community-hospital joint management for patients, and to provide follow-up online or offline every 3 months lasting for 10 years. Mainly, the objective of this study is to observe the blood glucose control outcome of T1DM patients. Secondly, the control of comprehensive metabolic indicators such as blood pressure and blood lipid, occurrence and progression of acute and chronic complications, and psychosocial status were included as well, expecting to provide scientific evidence for continuously improving the quality of T1DM management.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 years old;
* Diagnosed as type 1 diabetes according to World Health Organization (WHO) criteria in 1999;
* Be able to use smart mobile phones;
* Informed consent and voluntary participation.

Exclusion Criteria:

* Secondary diabetes;
* Complicated with malignant diseases, such as cancer, hepatic and renal failure;
* Complicated with cognitive impairment or mental illness;
* Be pregnant or lactating at the time of enrollment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 1 diabetes from in-patient and out-patient.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2032-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Outcome evaluation at 10 years.
  HbA1c is one of the indicators that reflects the level of blood glucose control overall. Blood sample will be required and tested.
Time in range (TIR) | Outcome evaluation at 10 years.
  TIR is one of the indicators that reflects the level of blood glucose control from the point of view of target time. Continuous glucose monitoring (CGM) devices will be used.
Incidence of hypoglycemia | Outcome evaluation at 10 years.
  Incidence of hypoglycemia is one of the indicators that reflects the level of blood glucose control. Hypoglycemia is defined as blood glucose lower than 3.9mmol/L with or without symptoms. Incidence of hypoglycemia is occurence times per month according to patients self-reported.

SECONDARY OUTCOMES:
Comprehensive metabolic control | Outcome evaluation at 10 years.
  Blood pressure is one of the control level comprehensive metabolic indicators, including systolic blood pressure (SBP) and diastolic blood pressure (DBP).
Comprehensive metabolic control | Outcome evaluation at 10 years.
  Blood lipid is one of the control level of comprehensive metabolic indicators, including total cholesterol (TC), total triglyceride (TG), high-density lipoprotein cholesterol (HDL-C) and low-density lipoprotein cholesterol (LDL-C).
Occurrence of Diabetes-related complications. | Outcome evaluation at 10 years.
  To observe and analyze occurrence of diabetes-related acute and chronic complications. Acute complications of diabetes include diabetic ketoacidosis (DKA), hypoglycemia and Hyperglycemic Hyperosmolar Syndrome (HHS). Chronic complications of diabetes including retinopathy, neuropathy nephropathy and lower extremity amputations (LEA). Other diabetes-related complications include cardiovascular disease, heart failure, stroke and death.
Progression of Diabetes-related complications. | Outcome evaluation at 10 years.
  To observe and analyze progression of diabetes-related acute and chronic complications. Acute complications of diabetes include diabetic ketoacidosis (DKA), hypoglycemia and Hyperglycemic Hyperosmolar Syndrome (HHS). Chronic complications of diabetes including retinopathy, neuropathy nephropathy and lower extremity amputations (LEA). Other diabetes-related complications include cardiovascular disease, heart failure, stroke and death.
Anxiety condition. | Outcome evaluation at 10 years.
  Anxiety condition is one of the psychosocial status indicators, and Self-Rating Anxiety Scale (SAS) will be used to assess anxiety level. The score ranges from 20 to 100, and higher score indicates more prone to anxiety.
Anxiety condition. | Outcome evaluation at 10 years.
  Anxiety condition is one of the psychosocial status indicators. Generalized Anxiety Disorder 7-Item Scale (GAD-7 scale) will be used to assess anxiety symptoms. The score ranges from 0 to 7, and higher score indicates more anxiety symptoms.
Depression condition. | Outcome evaluation at 10 years.
  Depression condition is one of the psychosocial status indicators, and Self-Rating Depression Scale (SDS) will be used to assess depression level. The level of depression is measured by depression severity index. The index ranges from 0.25 to 1.0, with higher scores associated with greater depression.
Depression condition. | Outcome evaluation at 10 years.
  Depression condition is one of the psychosocial status indicators, and Patient Health Questionnaire-9 (PHQ-9) will be used to assess depression level. The score ranges from 0 to 27. A higher score indicates a higher degree of depression.
Depression condition. | Outcome evaluation at 10 years.
  Depression condition is one of the psychosocial status indicators, and Problem Areas in Diabetes-Short form (PAID-5) will be used to evaluate the diabetes related emotional distress, which is strongly association with depression. A score ≥40 indicates high diabetes-related distress.
Life quality. | Outcome evaluation at 10 years.
  Life quality is one of the psychosocial status indicators, and specific scales as World Health Organization-5 well-being index (WHO-5) will be used to assess this factor. A score <50 indicates poor psychological well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yang, PhD, Study Director — Peking University Third Hospital; Kun Yang, MD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China